CLINICAL TRIAL: NCT03179839
Title: The Study of Mindfulness Based Cognitive Therapy and Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBCT2017
Record Dates: First submitted 2017-05-14; First posted 2017-06-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Mindfulness-Based Cognitive Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Mindfulness-Based Cognitive Therapy; Sertraline; Fluvoxamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based Cognitive Therapy (Experimental): MBCT group is a treatment group used mindfulness-based cognitive therapy, and guided by two therapists for 10 sessions. Every collection of about 6-8 patients is a closed structural group. Each session lasts 2.5 hours once a week, and has daily homework assignments.
  Interventions: Behavioral: Mindfulness-based Cognitive Therapy
- Psycho-education Program (Placebo Comparator): The program is consists of the information and principle of treatment for OCD, group sharing, supporting and discussion.
  Interventions: Behavioral: Psycho-education Program
- SSRIs Therapy (Active Comparator): This is a control group that can choose to use SSRI drugs which the SFDA approved for the treatment of OCD (Sertraline, Fluvoxamine, initial dose of 50 mg).
  Interventions: Drug: sertraline, fluvoxamine

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Therapy — The intervention will be carried out according to the handbook of the Dr. Didonna. There is a Session Agenda from Dr. Didonna for the use of the Instructor and session handouts for the participants. Some records of mindfulness practices will be given to participants for facilitating practice between sessions. Before each session, the instructor needs to review the session agenda and prepare copies of handouts for participants.
  MBCT instructors were experienced psychotherapists and psychiatrists with several years' expertise in OCD treatment. They had been trained by one of the founders of MBCT, Mark Williams and the founder of MBCT for OCD, Fabrizio Didonna. Supervision will be provided by Dr.Didonna.
  Arms: Mindfulness-based Cognitive Therapy
Behavioral: Psycho-education Program — As a widely used placebo control condition, the Psycho-Education Program can play an active role through the psychological suggestion and forward thinking mostly. It is designed to be similar with MBCT in level of structure, setting and other non-specific effects of psychological intervention. All instructors will be qualified graduate students who major in clinical psychology with training in cognitive behavioral therapy and psychodynamic therapy.
  Arms: Psycho-education Program
Drug: sertraline, fluvoxamine — The participants can be adjustable once a week dose and the maximum dose does not exceed the maximum amount of instructions. And benzodiazepine drugs also can be used by the OCD patients with sleep disorders, but not be used continuously for more than two weeks. Besides this, other psychotropic drugs are not allowed to use. The use of drugs in this study are commonly used drugs with good safety, and its common adverse reactions include dry mouth, constipation, nausea, indigestion, dizziness, fatigue, sweating and so on.
  Arms: SSRIs Therapy

SUMMARY:
The primary objective of the study is to evaluate the clinical curative effect of MBCT to reduce obsessive and compulsive symptoms. Moreover, the investigators will also explore a MBCT manual for Chinese patients with OCD, which can be widely applied to the clinical practice.

There are two parts of the study. The first part is a qualitative research with two pilot MBCT groups. The second part of this study is a single-blind randomized controlled trial with three study arms: one - third of participants receive group mindfulness-based cognitive therapy led by trained MBCT psychotherapists or psychiatrists in addition to medication, one - third of participants receive group psycho-education program and one - third of participants receive drug therapy as usual. All participants have 10 sessions intervention and assessments.

DETAILED DESCRIPTION:
The qualitative research will use grounded theory path to interview therapists and patients for 60 minutes in the baseline, after 5 weeks treatments and after the 10 weeks treatments. The subjective experience of the therapists and patients in two pilot MBCT groups will be described and explained. And the entire process of treatments will be participatory observed.

In the second part of the study, all patients will take blood test and functional magnetic resonance imaging (fMRI) scan in the baseline and after 10 weeks, to gather data in genetics and imaging features, which can help the study to discover biological indicators of the curative effect. And after the patients and their custodians signed the consent form, all of participants will be blindly assigned to three groups by a predetermined random table which is generated by Microsoft Excel 2010 for ensuring randomly fair distribution across conditions. The investigators will not decode these numbers until the intervention group is assigned.

As the research tools, a range of self-rating scales, other-rating scales and behavioral and physiological measures will be mainly applied to assess clinical symptoms of participants at baseline (week 0), mid-treatment (week 4), at the end of acute treatment (week 10), and during the maintenance phase (week 14, 22 and 34).

After 10 sessions, all the participants including the non-responders and the responders (ie, decrease in Yale-Brown Obsessive Compulsive Scale [YBOCS] scores ≥ 25%) will enter the maintenance phase for 6 months. The participants in MBCT group will continue MBCT treatments at home. The participants in drug therapy group will continue on their treatment program without changing the type and dosage of medication they have been using. By comparing clinical symptoms, such as obsessive and compulsive symptoms, anxiety, depression, quality of life and other clinical symptoms and behavior, the study will describe the short-term and long-term effects of MBCT in patients with DSM-IV obsessive-compulsive disorder (OCD).

ELIGIBILITY:
Inclusion Criteria:

* Participants should suffer from clinically OCD symptoms and have a DSM-IV Axis Ⅰ diagnosis of OCD (M.I.N.I.)
* 12≤ Y-BOCS score ≤25
* Male or female, 18 years old to 54 years of age
* Junior middle school education or above
* Have not yet accepted psychiatric medication, or had received irregular medication treatment and have been discontinued 8 weeks
* Have enough visual and acoustic ability to complete the inspection required for the study
* Each patient and his guardian must understand the nature of this study and sign the informed consent form

Exclusion Criteria:

* meet DSM-IV Axis Ⅰ diagnostic criteria for other psychiatric disorders
* persons with severe physical disease or central nervous system disease
* have a strong negative concept or a high risk of suicide
* substance abuse, pregnancy or the preparation of recently pregnant women and lactating women
* severe obsessive compulsive symptoms, so that patients can not complete the required assessment and treatment intervention
* at the same time to accept MECT or other psychological therapy
* patients had previously received treatment of mindfulness-based intervention, and no significant effect

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale | Change from baseline up to week 34
  Yale-Brown Obsessive-Compulsive Scale is a medical semi-structured questionnaire with a total of 10 items that measure the severity of Obsessive thinking and compulsive behavior on a scale of 0 = None; 1 = Sub-threshold; 2 =Mild; 3 =Moderate; and 4 = Severe. The total score is to be got by adding every score of all the items. And the higher the score is, the more severe OC symptoms are.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale | Change from baseline up to week 34
  Hamilton Anxiety Scale is the most common other-rating scale for clinical assessment of anxiety status and suitable for adults with anxiety symptoms. There are 14 items with each symptom rated on a five-point Scale.
Hamilton Depression Scale-24 | Change from baseline up to week 34
  Hamilton Depression Scale-24 is the most common other-rating scale for clinically assessing the state of depression and suitable for adults with depressive symptoms. There are 24 items rated to each symptom and most of the items used 0 to 4 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Shen, Senior, Study Director — Shanghai Mental Health Center
Locations (1):
- Clinical psychiatrist, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No